CLINICAL TRIAL: NCT06900556
Title: Effect of Post-exercise Dry Cupping Therapy on Muscle Recovery
Brief Title: Dry Cupping for Recovery From Muscle Damage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024_25_04
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Muscle Damage
MeSH Terms: interventions — Suction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry cupping with suction (Experimental)
  Interventions: Procedure: Dry cupping with suction
- Dry cupping without suction (Sham Comparator)
  Interventions: Procedure: Dry cupping without suction

INTERVENTIONS:
Procedure: Dry cupping with suction — Dry cupping with suction applied to the biceps
  Arms: Dry cupping with suction
Procedure: Dry cupping without suction — Dry cupping without suction applied to the biceps
  Arms: Dry cupping without suction

SUMMARY:
This study compares the effect of dry cupping to placebo cupping after muscle-damaging exercise on recovery of muscle strength, muscle swelling, and muscle soreness.

DETAILED DESCRIPTION:
Dry cupping is a technique where cups are placed on the skin and a suction device is used to remove air from the cups. This study aims to investigate whether dry cupping therapy can enhance muscle recovery following exercise by measuring muscle soreness, swelling, and strength in the biceps. Six sets of biceps curls (emphasizing concentric and eccentric overload) will be performed on each arm, followed by dry cupping with suction applied to one arm (experimental) and dry cupping without suction (placebo) applied to the opposite arm. Experimental and placebo arms for each participant will be randomized. Before exercise and immediately, 24 hours, 48 hours, and 72 hours after exercise, muscle strength, muscle swelling (ultrasound), and muscle soreness (visual analog scale) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-35 years old
* Experienced with upper arm resistance training for at least 3 months

Exclusion Criteria:

* Conditions that might make exercise dangerous (determined by "yes" answers to the "Get Active Questionnaire")
* Open wounds, scars, eczema, or other skin sensitivities on the biceps area

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Biceps isometric strength measured by dynamometry (Nm) | Change over 72 hours

SECONDARY OUTCOMES:
Biceps swelling (muscle thickness) measured with ultrasound (cm) | Change over 24 hours
Biceps muscle soreness measured with a visual analog scale from 0 (no soreness) to 10 (maximal soreness) | Change over 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No